CLINICAL TRIAL: NCT06073990
Title: A Quasi-experimental Study Design of Evaluation the Effects of Brief Behavioral Therapy for Insomnia on Regulating Stress and Sleep Quality in Middle-aged and Older Adults With Chronic Insomnia
Brief Title: Brief Behavioral Therapy for Insomnia(BBTi) in Middle-aged and Older Adults With Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-112-175
Record Dates: First submitted 2023-08-23; First posted 2023-10-10 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-07

CONDITIONS: Chronic Insomnia; Older Adults; Sleep Hygiene
Keywords: Brief Behavioral Treatment for Insomnia; Chronic Insomnia; Older adults; Sleep Hygiene
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brief Behavioral Treatment for Insomnia (BBTi) (Experimental): In the post-intervention group, the investigators collected data at the 1-week, 2-week, and 3-week marks following the intervention.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTi)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia (BBTi) — The intervention consists of four weeks of BBTi. During the first week, participants will receive face-to-face sleep assessments and sleep hygiene education. In the second week, a phone interview will be conducted to assess the patient's progress and provide appropriate relaxation techniques. Unsatisfactory responses to sleep restriction therapy or stimulation control methods will be addressed through face-to-face interviews in the third week. The fourth week will involve an overall review and evaluation conducted via a telephone interview.

SUMMARY:
This study aims to investigate whether a four-week BBTi program can effectively improve chronic insomnia and reduce overall stress in middle-aged and elderly individuals.

DETAILED DESCRIPTION:
This study will be conducted a single-group pre-test and post-test design, aiming to recruit 80 subjects who will undergo a four-week BBTi intervention. Participants will be selected from sleep counseling patients referred by sleep specialists. Inclusion criteria include: 1) individuals aged 40 years and above; 2) experiencing sleep disturbances; 3) willing to participate in the research project and provide informed consent. Cognitive impairment will exclude. The intervention consists of four weeks of BBTi. During the first week, participants will receive face-to-face sleep assessments and sleep hygiene education. In the second week, a phone interview will be conducted to assess the patient's progress and provide appropriate relaxation techniques. Unsatisfactory responses to sleep restriction therapy or stimulation control methods will be addressed through face-to-face interviews in the third week. The fourth week will involve an overall review and evaluation conducted via a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 40 years and above,
* experiencing sleep disturbances,
* willing to participate in the research project and provide informed consent

Exclusion Criteria:

●Cognitive impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity (T1) | the first week
  The investigators collected the insomnia severity from participants:
  The Insomnia Severity Scale (ISI) comprises seven items. Each question is scored on a scale of 0 to 4 points, and total scores are ranged 0-28 points. A higher total score indicates a higher severity of insomnia. Specifically, a score ranging from 0 to 7 indicates no significant insomnia issues, while a score of 8 to 14 signifies mild sleep difficulties. An ISI score falling within the range of 15 to 21 reflects moderate insomnia, and a score of 22 to 28 indicates severe insomnia.
Insomnia severity (T2) | the second week
  The investigators collected the insomnia severity from participants:
  The Insomnia Severity Scale (ISI) comprises seven items. Each question is scored on a scale of 0 to 4 points, and total scores are ranged 0-28 points. A higher total score indicates a higher severity of insomnia. Specifically, a score ranging from 0 to 7 indicates no significant insomnia issues, while a score of 8 to 14 signifies mild sleep difficulties. An ISI score falling within the range of 15 to 21 reflects moderate insomnia, and a score of 22 to 28 indicates severe insomnia.
Insomnia severity (T3) | the third week
  The investigators collected the insomnia severity from participants:
  The Insomnia Severity Scale (ISI) comprises seven items. Each question is scored on a scale of 0 to 4 points, and total scores are ranged 0-28 points. A higher total score indicates a higher severity of insomnia. Specifically, a score ranging from 0 to 7 indicates no significant insomnia issues, while a score of 8 to 14 signifies mild sleep difficulties. An ISI score falling within the range of 15 to 21 reflects moderate insomnia, and a score of 22 to 28 indicates severe insomnia.
Insomnia severity (T4) | the fourth week
  The investigators collected the insomnia severity from participants:
  The Insomnia Severity Scale (ISI) comprises seven items. Each question is scored on a scale of 0 to 4 points, and total scores are ranged 0-28 points. A higher total score indicates a higher severity of insomnia. Specifically, a score ranging from 0 to 7 indicates no significant insomnia issues, while a score of 8 to 14 signifies mild sleep difficulties. An ISI score falling within the range of 15 to 21 reflects moderate insomnia, and a score of 22 to 28 indicates severe insomnia.
Sleep health (T1) | the first week
  The researchers collected data using the Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) questionnaire from the participants.
  The RU-SATED questionnaire consists of six questions, each evaluating distinct facets of sleep health. These questions encompass aspects such as sleep regularity, sleep satisfaction, daytime alertness, sleep timing, sleep efficiency, and sleep duration. Each question is rated on a scale of 0 to 2 points, resulting in a total score that ranges from 0 to 12 points. A higher total score across these six questions indicates a greater level of sleep health.
Sleep health (T2) | the second week
  The researchers collected data using the Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) questionnaire from the participants.
  The RU-SATED questionnaire consists of six questions, each evaluating distinct facets of sleep health. These questions encompass aspects such as sleep regularity, sleep satisfaction, daytime alertness, sleep timing, sleep efficiency, and sleep duration. Each question is rated on a scale of 0 to 2 points, resulting in a total score that ranges from 0 to 12 points. A higher total score across these six questions indicates a greater level of sleep health.
Sleep health (T3) | the third week
  The researchers collected data using the Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) questionnaire from the participants.
  The RU-SATED questionnaire consists of six questions, each evaluating distinct facets of sleep health. These questions encompass aspects such as sleep regularity, sleep satisfaction, daytime alertness, sleep timing, sleep efficiency, and sleep duration. Each question is rated on a scale of 0 to 2 points, resulting in a total score that ranges from 0 to 12 points. A higher total score across these six questions indicates a greater level of sleep health.
Sleep health (T4) | the fourth week
  The researchers collected data using the Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) questionnaire from the participants.
  The RU-SATED questionnaire consists of six questions, each evaluating distinct facets of sleep health. These questions encompass aspects such as sleep regularity, sleep satisfaction, daytime alertness, sleep timing, sleep efficiency, and sleep duration. Each question is rated on a scale of 0 to 2 points, resulting in a total score that ranges from 0 to 12 points. A higher total score across these six questions indicates a greater level of sleep health.
Sleep Diary_Sleep efficacy (%) (T1) | the first week
  The researchers obtained sleep diaries from the participants.
  The sleep diary is a subjective record in which subjects document their sleep patterns. The following aspects can be assessed through the sleep diary:
  Total Sleep Time (TST):Calculated as the time elapsed from the moment of waking to the time of falling asleep.
  Sleep Efficiency: The ratio of total sleep time (TST) to time in bed (TIB) (multiplied by 100 to yield a percentage)
Sleep Diary_Sleep efficacy (%) (T2) | the second week
  The researchers obtained sleep diaries from the participants.
  The sleep diary is a subjective record in which subjects document their sleep patterns. The following aspects can be assessed through the sleep diary:
  Total Sleep Time (TST):Calculated as the time elapsed from the moment of waking to the time of falling asleep.
  Sleep Efficiency: The ratio of total sleep time (TST) to time in bed (TIB) (multiplied by 100 to yield a percentage)
Sleep Diary_Sleep efficacy (%) (T3) | the third week
  The researchers obtained sleep diaries from the participants.
  The sleep diary is a subjective record in which subjects document their sleep patterns. The following aspects can be assessed through the sleep diary:
  Total Sleep Time (TST):Calculated as the time elapsed from the moment of waking to the time of falling asleep.
  Sleep Efficiency: The ratio of total sleep time (TST) to time in bed (TIB) (multiplied by 100 to yield a percentage)
Sleep Diary_Sleep efficacy (%) (T4) | the fourth week
  The researchers obtained sleep diaries from the participants.
  The sleep diary is a subjective record in which subjects document their sleep patterns. The following aspects can be assessed through the sleep diary:
  Total Sleep Time (TST):Calculated as the time elapsed from the moment of waking to the time of falling asleep.
  Sleep Efficiency: The ratio of total sleep time (TST) to time in bed (TIB) (multiplied by 100 to yield a percentage)
Anxiety (T1) | the first week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of anxiety. A score falling between 8 and 10 suggests possible anxiety. A score exceeding 11 indicates the presence of anxiety in the patient.
Anxiety (T2) | the second week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of anxiety. A score falling between 8 and 10 suggests possible anxiety. A score exceeding 11 indicates the presence of anxiety in the patient.
Anxiety (T3) | the third week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of anxiety. A score falling between 8 and 10 suggests possible anxiety. A score exceeding 11 indicates the presence of anxiety in the patient.
Anxiety (T4) | the fourth week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of anxiety. A score falling between 8 and 10 suggests possible anxiety. A score exceeding 11 indicates the presence of anxiety in the patient.
Depression (T1) | the first week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of depression. A score falling between 8 and 10 suggests possible depression. A score exceeding 11 indicates the presence of depression in the patient.
Depression (T2) | the second week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of depression. A score falling between 8 and 10 suggests possible depression. A score exceeding 11 indicates the presence of depression in the patient.
Depression (T3) | the third week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of depression. A score falling between 8 and 10 suggests possible depression. A score exceeding 11 indicates the presence of depression in the patient.
Depression (T4) | the fourth week
  The researchers collected data using the Hospital Anxiety and Depression Scale (HADS) from the participants.
  This scale, originally developed by Zigmond and Snaith in 1983, was designed for individuals with physical illnesses. It consists of a total of 14 items, each scored on a four-point scale (ranging from 0 to 3 points). The scale comprises 7 items related to anxiety and 7 items related to depression. Interpretation of the scores is as follows:
  A total score of less than 8 indicates the absence of depression. A score falling between 8 and 10 suggests possible depression. A score exceeding 11 indicates the presence of depression in the patient.
Stress index (ms2) (T1) | the first week
  The investigators use EUREKA to detect the heartbeat variation of participants and analyze the pressure index.
  Stress index (ms2) < 50: abnormal records; 50-150: Normal; 150-500: fatigue state or greater physical and mental stress; 500-900: severe physical and mental stress; > 900 extreme physical and mental stress or other physical diseases.
Stress index (ms2) (T3) | the third week
  The investigators use EUREKA to detect the heartbeat variation of participants and analyze the pressure index.
  Stress index (ms2) < 50: abnormal records; 50-150: Normal; 150-500: fatigue state or greater physical and mental stress; 500-900: severe physical and mental stress; > 900 extreme physical and mental stress or other physical diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No